CLINICAL TRIAL: NCT00093015
Title: Trial to Reduce Cardiovascular Events With Aranesp® Therapy
Brief Title: Trial to Reduce Cardiovascular Events With Aranesp® Therapy (TREAT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20010184; TREAT
Record Dates: First submitted 2004-09-28; First posted 2004-09-29 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Kidney Disease; Diabetes Mellitus; Anemia
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: darbepoetin alfa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Volume and dose frequency changes resembling dosing in the active treatment group
  Arms: Placebo
Drug: darbepoetin alfa — Starting dose : 0.75 mcg/kg subcutaneous (SC) every two weeks (Q2W); subsequent doses titrated to achieve hemoglobin (Hb) target of 13.0 g/dL
  Arms: Active

SUMMARY:
The purpose of this study is to assess the impact of treatment of anemia with darbepoetin alfa to a hemoglobin target of 13 g/dL on (1) all-cause mortality and nonfatal cardiovascular events, and (2) progression to end-stage renal disease or death, in subjects with chronic kidney disease and type 2 diabetes mellitus.

Academic PI/Executive Committee Chairman: Marc Pfeffer, MD, PhD

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin less than or equal to 11 g/dL
* History of Chronic Kidney Disease
* eGFR (estimated glomerular filtration rate) greater than or equal to 20 mL/min/1.73 m2 and less than or equal to 60 mL/min/1.73 m2
* Tsat (transferrin saturation) greater than 15%

Exclusion Criteria:

* Uncontrolled hypertension
* Erythropoietic protein use within 12 weeks of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4038 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Lewis EF, Pfeffer MA, Feng A, Uno H, McMurray JJ, Toto R, Gandra SR, Solomon SD, Moustafa M, Macdougall IC, Locatelli F, Parfrey PS; TREAT Investigators. Darbepoetin alfa impact on health status in diabetes patients with kidney disease: a randomized trial. Clin J Am Soc Nephrol. 2011 Apr;6(4):845-55. doi: 10.2215/CJN.06450710. Epub 2011 Jan 6. PMID 21212421
- [Background] McMurray JJ, Uno H, Jarolim P, Desai AS, de Zeeuw D, Eckardt KU, Ivanovich P, Levey AS, Lewis EF, McGill JB, Parfrey P, Parving HH, Toto RM, Solomon SD, Pfeffer MA. Predictors of fatal and nonfatal cardiovascular events in patients with type 2 diabetes mellitus, chronic kidney disease, and anemia: an analysis of the Trial to Reduce cardiovascular Events with Aranesp (darbepoetin-alfa) Therapy (TREAT). Am Heart J. 2011 Oct;162(4):748-755.e3. doi: 10.1016/j.ahj.2011.07.016. PMID 21982669
- [Background] Mix TC, Brenner RM, Cooper ME, de Zeeuw D, Ivanovich P, Levey AS, McGill JB, McMurray JJ, Parfrey PS, Parving HH, Pereira BJ, Remuzzi G, Singh AK, Solomon SD, Stehman-Breen C, Toto RD, Pfeffer MA. Rationale--Trial to Reduce Cardiovascular Events with Aranesp Therapy (TREAT): evolving the management of cardiovascular risk in patients with chronic kidney disease. Am Heart J. 2005 Mar;149(3):408-13. doi: 10.1016/j.ahj.2004.09.047. PMID 15864229
- [Background] Pfeffer MA, Burdmann EA, Chen CY, Cooper ME, de Zeeuw D, Eckardt KU, Feyzi JM, Ivanovich P, Kewalramani R, Levey AS, Lewis EF, McGill JB, McMurray JJ, Parfrey P, Parving HH, Remuzzi G, Singh AK, Solomon SD, Toto R; TREAT Investigators. A trial of darbepoetin alfa in type 2 diabetes and chronic kidney disease. N Engl J Med. 2009 Nov 19;361(21):2019-32. doi: 10.1056/NEJMoa0907845. Epub 2009 Oct 30. PMID 19880844
- [Background] Solomon SD, Uno H, Lewis EF, Eckardt KU, Lin J, Burdmann EA, de Zeeuw D, Ivanovich P, Levey AS, Parfrey P, Remuzzi G, Singh AK, Toto R, Huang F, Rossert J, McMurray JJ, Pfeffer MA; Trial to Reduce Cardiovascular Events with Aranesp Therapy (TREAT) Investigators. Erythropoietic response and outcomes in kidney disease and type 2 diabetes. N Engl J Med. 2010 Sep 16;363(12):1146-55. doi: 10.1056/NEJMoa1005109. PMID 20843249
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Lewis EF, Claggett B, Parfrey PS, Burdmann EA, McMurray JJ, Solomon SD, Levey AS, Ivanovich P, Eckardt KU, Kewalramani R, Toto R, Pfeffer MA. Race and ethnicity influences on cardiovascular and renal events in patients with diabetes mellitus. Am Heart J. 2015 Aug;170(2):322-9. doi: 10.1016/j.ahj.2015.05.008. Epub 2015 May 22. PMID 26299230
- [Derived] Bello NA, Pfeffer MA, Skali H, McGill JB, Rossert J, Olson KA, Weinrauch L, Cooper ME, de Zeeuw D, Rossing P, McMurray JJ, Solomon SD. Retinopathy and clinical outcomes in patients with type 2 diabetes mellitus, chronic kidney disease, and anemia. BMJ Open Diabetes Res Care. 2014 Apr 6;2(1):e000011. doi: 10.1136/bmjdrc-2013-000011. eCollection 2014. PMID 25452859
- [Derived] Skali H, Parving HH, Parfrey PS, Burdmann EA, Lewis EF, Ivanovich P, Keithi-Reddy SR, McGill JB, McMurray JJ, Singh AK, Solomon SD, Uno H, Pfeffer MA; TREAT Investigators. Stroke in patients with type 2 diabetes mellitus, chronic kidney disease, and anemia treated with Darbepoetin Alfa: the trial to reduce cardiovascular events with Aranesp therapy (TREAT) experience. Circulation. 2011 Dec 20;124(25):2903-8. doi: 10.1161/CIRCULATIONAHA.111.030411. Epub 2011 Nov 21. PMID 22104547
- [Derived] Pfeffer MA, Burdmann EA, Chen CY, Cooper ME, de Zeeuw D, Eckardt KU, Ivanovich P, Kewalramani R, Levey AS, Lewis EF, McGill J, McMurray JJ, Parfrey P, Parving HH, Remuzzi G, Singh AK, Solomon SD, Toto R, Uno H; TREAT Investigators. Baseline characteristics in the Trial to Reduce Cardiovascular Events With Aranesp Therapy (TREAT). Am J Kidney Dis. 2009 Jul;54(1):59-69. doi: 10.1053/j.ajkd.2009.04.008. Epub 2009 Jun 5. PMID 19501439
- [Derived] Pfeffer MA; TREAT Executive Committee. An ongoing study of anemia correction in chronic kidney disease. N Engl J Med. 2007 Mar 1;356(9):959-61. doi: 10.1056/NEJMc066568. No abstract available. PMID 17329707
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 25 Aug 2004 Last Subject Enrolled: 04 Dec 2007
Groups:
- Placebo: Subcutaneous placebo when hemoglobin concentration was ≥ 9.0 g/dL. Received subcutaneous rescue therapy (once monthly) with darbepoetin alfa in a blinded fashion if the hemoglobin concentration was <9.0 g/dL until the hemoglobin concentration was ≥ 9.0 g/dL.
- Darbepoetin Alfa: Subcutaneous darbepoetin alfa at a starting dose of 75 mcg/kg once every 2 weeks, titrated to maintain a hemoglobin concentration of 13.0 g/dL. Dosing was switched to once monthly when two consecutive hemoglobin concentrations between 12.0 and 13.5 g/dL were observed.
Period: Overall Study
Arm/Group | Placebo | Darbepoetin Alfa
Started | 2026 | 2012
Received Study Medication | 2019 | 2004
Completed | 1361 | 1348
Not Completed | 665 | 664
Not completed — Withdrawal by Subject | 194 | 171
Not completed — Lost to Follow-up | 96 | 108
Not completed — Death | 375 | 385

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa | Placebo | Total
Number analyzed (Participants) | 2012 | 2026 | 4038
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (10.7) | 67.5 (10.6) | 67.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1178 | 1134 | 2312
  Male | 834 | 892 | 1726
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 1270 | 1300 | 2570
  Black or African American | 414 | 401 | 815
  Hispanic or Latino | 273 | 265 | 538
  Asian | 35 | 43 | 78
  Japanese | 8 | 3 | 11
  American Indian or Alaska Native | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Aborigine | 2 | 1 | 3
  Other | 5 | 4 | 9
History of cardiovascular disease [Number; unit: Participant] — Cardiovascular disease history is based on the cardiovascular medical history case report form.
  Participant
    With history of cardiovascular disease | 1287 | 1355 | 2642
    Without history of cardiovascular disease | 725 | 671 | 1396
Baseline proteinuria level [Number; unit: Participants] — Baseline proteinuria level (g/g creat). Baseline proteinuria is defined as the last non-missing measurement prior or on the day of first investigational product.
  Participants
    >= 1 g/g creat | 686 | 711 | 1397
    < 1 g/g creat | 1324 | 1315 | 2639

OUTCOME MEASURES:

1. Primary Outcome: Time to All-cause Mortality or Cardiovascular (CV) Events Including Hospitalization Due to Acute Myocardial Ischemia, Congestive Heart Failure (CHF), Myocardial Infarction (MI), and Cerebrovascular Accident (CVA)
Description: Time from randomization to the first confirmed composite event. Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: Until a primary cardiovascular event (death, myocardial ischemia, congestive heart failure, myocardial infarction or cerebrovascular accident) occurred or 28 March 2009, whichever occurred first
Population: The analysis followed intent-to-treat principles. Subjects were analyzed as randomized using all available follow-up information.
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 602 | 632
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.41, Log Rank — Nominal p-value from a 2-sided log rank test is presented. The primary cardiovascular composite endpoint was tested at the 0.04056 significance level at final analysis after accounting for 4 planned interim analyses (overall alpha = 0.048); A 2-sided log-rank test comparing the survival functions of the 2 groups stratified by baseline proteinuria and CV disease (CVD) history; Cox Proportional Hazard = 1.05, 95% CI [0.94 to 1.17] — Treatment effect was estimated using a hazards ratio and 95% confidence interval (CI) obtained from a Cox proportional hazards model stratified by baseline proteinuria and CVD history. Hazard ratio (darbepoetin alfa / placebo)

2. Primary Outcome: Time to All-cause Mortality or End Stage Renal Disease (ESRD)
Description: Time from randomization to first event of all-cause mortality or ESRD. Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 618 | 652
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.29, Log Rank — Nominal p-value from a 2-sided log rank test is presented. The primary renal composite endpoint was tested at the 0.002 significance level at final analysis; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.06, 95% CI [0.95 to 1.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to All-cause Mortality
Description: Time from randomization to all-cause mortality. Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 395 | 412
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.48, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.05, 95% CI [0.92 to 1.21] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Cardiovascular Mortality
Description: Time from randomization to cardiovascular (CV) mortality. Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 250 | 259
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.61, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.05, 95% CI [0.88 to 1.25] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Myocardial Infarction
Description: Time from randomization to fatal or non-fatal myocardial infarction (MI). Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 129 | 124
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.73, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.96, 95% CI [0.75 to 1.23] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Cerebrovascular Accident
Description: Time from randomization to fatal or non-fatal cerebrovascular accident (CVA). Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 53 | 101
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p < 0.001, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.92, 95% CI [1.38 to 2.68] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Congestive Heart Failure
Description: Time from randomization to fatal or non-fatal congestive heart failure(CHF). Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 229 | 205
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.24, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.89, 95% CI [0.74 to 1.08] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to End Stage Renal Disease
Description: Time from randomization to end stage renal disease (ESRD). Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 330 | 338
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.83, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.02, 95% CI [0.87 to 1.18] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Rate of Decline in Estimated Glomerular Filtration Rate (eGFR) Relative to Baseline
Description: GFR was estimated using the following MDRD formula: 186 x [Serum creatinine]^(-1.154) x [Age]^(-0.203) x [0.742 if subject is female] x [1.210 if subject is black]. Change from baseline in eGFR at week 49 for each treatment group are presented. The treatment effect of the rate of decline in eGFR per year was estimated using the mixed model.
Time Frame: as for outcome 1
Population: Subjects were analyzed as randomized using all available eGFR measurements, except eGFR measurements measured after subjects develop ESRD since creatinine measurements were no longer reliable or meaningful for eGFR calculation.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
mL/min/1.73m^2 | -1.89 (10.60) | -1.30 (10.81)
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis — Nominal p-value is from the term treatment group*visit in the mixed model; Adjusted for baseline eGFR and the stratification factors of proteinuria and CVD history; Slope = -0.12, 95% CI [-0.51 to 0.26] — Estimated difference in rate of decline in eGFR per year between darbepoetin alfa and placebo

10. Secondary Outcome: Change in Patient Reported Fatigue Relative to Baseline at Week 25
Description: Change in patient reported fatigue measured by the Functional Assessment of Cancer Therapy (FACT) - Fatigue scale from baseline to week 25. Range and direction of scale: 0 = most fatigue; 52 = least fatigue
Time Frame: Baseline and week 25
Population: Subjects with both the baseline and at least post-baseline measurement at week 25 for FACT-fatigue were included in the analysis and were analyzed as randomized. Last observation carried forward (LOCF) using last non-missing post-baseline value was used for missing post-baseline data for subjects who were still on study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 1769 | 1762
Units on a scale | 2.8 (10.3) | 4.2 (10.5)
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Nominal p-value is presented; Mean Difference (Final Values) = 1.33, 95% CI [0.64 to 2.02], Standard Deviation 0.35 — Difference (darbepoetin alfa - placebo)

11. Secondary Outcome: Time to Hospitalization Due to Acute Myocardial Ischemia
Description: Time from randomization to hospitalization due to acute myocardial ischemia. Kaplan-Meier estimate of the median time was not estimable due to low proportion of participants experiencing at least one events, therefore participants experiencing at least one event were summarized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 2026 | 2012
Participants | 49 | 41
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.40, Log Rank — Nominal p-value from a 2-sided log rank test is presented; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.84, 95% CI [0.55 to 1.27] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Differential follow-up up to 4.6 years
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 1219/2019 | 1235/2004
Other Adverse Events (participants affected / at risk) | 1547/2019 | 1571/2004
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2019) | Darbepoetin Alfa (N=2004)
Anaemia (Blood and lymphatic system disorders) | 155 | 65
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 2 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 2
Hypercoagulation (Blood and lymphatic system disorders) | 2 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 4
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
AV dissociation (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 17 | 18
Acute myocardial infarction (Cardiac disorders) | 28 | 33
Angina pectoris (Cardiac disorders) | 28 | 19
Angina unstable (Cardiac disorders) | 22 | 17
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 8 | 7
Arrhythmia supraventricular (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 3
Atrial fibrillation (Cardiac disorders) | 42 | 39
Atrial flutter (Cardiac disorders) | 5 | 6
Atrioventricular block (Cardiac disorders) | 3 | 2
Atrioventricular block complete (Cardiac disorders) | 8 | 7
Atrioventricular block second degree (Cardiac disorders) | 3 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 15 | 8
Cardiac arrest (Cardiac disorders) | 23 | 31
Cardiac disorder (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 40 | 38
Cardiac failure acute (Cardiac disorders) | 6 | 1
Cardiac failure chronic (Cardiac disorders) | 6 | 10
Cardiac failure congestive (Cardiac disorders) | 214 | 178
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 1
Cardiac valve sclerosis (Cardiac disorders) | 0 | 1
Cardiac valve vegetation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 19 | 17
Cardiogenic shock (Cardiac disorders) | 5 | 4
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 3 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 2
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 62 | 41
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 6 | 2
Diastolic dysfunction (Cardiac disorders) | 3 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 10 | 6
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Microvascular angina (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 63 | 78
Myocardial ischaemia (Cardiac disorders) | 18 | 10
Nodal arrhythmia (Cardiac disorders) | 1 | 2
Nodal rhythm (Cardiac disorders) | 1 | 0
Pacemaker generated arrhythmia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 4 | 1
Pericardial effusion (Cardiac disorders) | 3 | 2
Pericarditis (Cardiac disorders) | 2 | 2
Pleuropericarditis (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 7 | 5
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 1 | 1
Torsade de pointes (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 5 | 6
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Hypospadias (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Urachal abnormality (Congenital, familial and genetic disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Haematotympanum (Ear and labyrinth disorders) | 0 | 1
Otosalpingitis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Vestibular neuronitis (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 3
Cataract (Eye disorders) | 8 | 8
Cataract cortical (Eye disorders) | 0 | 1
Cataract diabetic (Eye disorders) | 2 | 0
Diabetic blindness (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 3 | 5
Eye haemorrhage (Eye disorders) | 3 | 3
Glaucoma (Eye disorders) | 2 | 0
Iridocyclitis (Eye disorders) | 0 | 1
Maculopathy (Eye disorders) | 1 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 3
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 16 | 14
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 2
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Bezoar (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 2
Colitis ischaemic (Gastrointestinal disorders) | 2 | 3
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic atony (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 2 | 6
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 | 1
Duodenitis (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 8 | 7
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 9 | 10
Gastritis erosive (Gastrointestinal disorders) | 1 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 28 | 21
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 10
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 3
Ileus (Gastrointestinal disorders) | 1 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 6
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 2
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Oesophageal polyp (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 5 | 8
Pancreatitis acute (Gastrointestinal disorders) | 4 | 5
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3
Volvulus (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 8 | 7
Adverse drug reaction (General disorders) | 4 | 7
Adverse event (General disorders) | 1 | 0
Asthenia (General disorders) | 9 | 9
Brain death (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 1
Catheter site inflammation (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 11 | 12
Death (General disorders) | 38 | 39
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 4
Generalised oedema (General disorders) | 4 | 3
Hernia (General disorders) | 0 | 1
Hernia obstructive (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Ischaemic ulcer (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 7 | 3
Necrobiosis (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 22 | 29
Oedema (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 7 | 6
Pain (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 3
Sudden cardiac death (General disorders) | 2 | 1
Sudden death (General disorders) | 11 | 12
Ulcer (General disorders) | 0 | 1
Wound necrosis (General disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 9 | 8
Cholecystitis acute (Hepatobiliary disorders) | 6 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 7 | 17
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 4
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 2
Sarcoidosis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 4
Abscess limb (Infections and infestations) | 5 | 3
Acute endocarditis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 4
Arteriovenous fistula site infection (Infections and infestations) | 1 | 2
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 2 | 3
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 4 | 3
Bacterial disease carrier (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 2 | 1
Breast cellulitis (Infections and infestations) | 0 | 2
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 20 | 32
Bronchitis bacterial (Infections and infestations) | 1 | 1
Bronchitis fungal (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 13 | 9
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 3
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 41 | 59
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Cervicitis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 3
Corynebacterium infection (Infections and infestations) | 1 | 0
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Dacryocystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Diabetic foot infection (Infections and infestations) | 8 | 11
Diabetic gangrene (Infections and infestations) | 0 | 4
Diarrhoea infectious (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 4 | 8
Embolic pneumonia (Infections and infestations) | 0 | 1
Emphysematous cystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 3
Encephalitis viral (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 3 | 3
Endocarditis bacterial (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Enterovirus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 3 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 11 | 19
Gas gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 27 | 31
Gastroenteritis viral (Infections and infestations) | 3 | 6
Gastrointestinal infection (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 2 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 5
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Infected bunion (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 5
Infection (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 0 | 5
Intervertebral discitis (Infections and infestations) | 2 | 2
Intraspinal abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 9 | 5
Localised infection (Infections and infestations) | 4 | 14
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 18 | 24
Osteomyelitis acute (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 2 | 3
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 1
Perirectal abscess (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 120 | 90
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 2 | 0
Post procedural infection (Infections and infestations) | 0 | 2
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 6
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 7
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 5 | 2
Pyelonephritis fungal (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 32 | 30
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 9 | 9
Sinusitis (Infections and infestations) | 2 | 6
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 3 | 3
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 3
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 2 | 0
Subacute endocarditis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 3 | 4
Tooth abscess (Infections and infestations) | 1 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 50 | 58
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 9 | 14
Uterine abscess (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 3
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 4
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 2
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 4
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Dialysis device complication (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 3
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Eyeball rupture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 5
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur fracture (Injury, poisoning and procedural complications) | 9 | 10
Fibula fracture (Injury, poisoning and procedural complications) | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 5 | 1
Heart injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 17 | 22
Humerus fracture (Injury, poisoning and procedural complications) | 8 | 4
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 2
Injury (Injury, poisoning and procedural complications) | 2 | 0
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 | 0
Intraocular lens dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 1
Joint sprain (Injury, poisoning and procedural complications) | 4 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 4
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 5
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 6
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 6
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 6 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Carotid bruit (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Medical observation (Investigations) | 0 | 1
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 40 | 29
Diabetes mellitus (Metabolism and nutrition disorders) | 30 | 24
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 22 | 26
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 5 | 12
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 6 | 9
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Enzyme abnormality (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 6 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 5 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 33
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 51 | 48
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 58 | 81
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 7
Hypovolaemia (Metabolism and nutrition disorders) | 5 | 5
Iron deficiency (Metabolism and nutrition disorders) | 1 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 1
Obesity (Metabolism and nutrition disorders) | 4 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 4
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 | 6
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 6
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 | 24
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 6
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1
Brain mass (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 11 | 8
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 3
Cerebral ischaemia (Nervous system disorders) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 37 | 72
Cerebrovascular disorder (Nervous system disorders) | 0 | 3
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 3 | 4
Dementia (Nervous system disorders) | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic coma (Nervous system disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 5 | 5
Dizziness (Nervous system disorders) | 3 | 5
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 3
Epilepsy (Nervous system disorders) | 0 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Global amnesia (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 3 | 5
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 3 | 5
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 4
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 2
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 4 | 6
Lacunar infarction (Nervous system disorders) | 1 | 5
Leukoaraiosis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 7
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 1
Sedation (Nervous system disorders) | 1 | 0
Senile dementia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 26 | 16
Syncope vasovagal (Nervous system disorders) | 3 | 3
Thalamic infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 18 | 28
Uraemic encephalopathy (Nervous system disorders) | 1 | 3
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Bipolar disorder (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 3 | 3
Conversion disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 5 | 7
Disorientation (Psychiatric disorders) | 0 | 1
Impaired self-care (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 4 | 3
Schizophrenia (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 3 | 1
Atonic urinary bladder (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 3 | 10
Bladder diverticulum (Renal and urinary disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 4 | 8
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Kidney enlargement (Renal and urinary disorders) | 1 | 0
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 6
Nephropathy (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 6 | 10
Neurogenic bladder (Renal and urinary disorders) | 2 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 2
Renal artery occlusion (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 4 | 3
Renal colic (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 3
Renal failure (Renal and urinary disorders) | 82 | 72
Renal failure acute (Renal and urinary disorders) | 69 | 70
Renal failure chronic (Renal and urinary disorders) | 180 | 223
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 6 | 11
Renal mass (Renal and urinary disorders) | 1 | 0
Renal papillary necrosis (Renal and urinary disorders) | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Stag horn calculus (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Breast calcifications (Reproductive system and breast disorders) | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 20 | 25
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 26 | 23
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin graft failure (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 | 20
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1
Abdominal cavity drainage (Surgical and medical procedures) | 1 | 0
Arteriovenous graft (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 0
Catheterisation cardiac (Surgical and medical procedures) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 1 | 0
Coronary revascularisation (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Leg amputation (Surgical and medical procedures) | 1 | 1
Limb operation (Surgical and medical procedures) | 1 | 0
Removal of inert matter from skin or subcutaneous tissue (Surgical and medical procedures) | 1 | 0
Skin graft (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 7 | 3
Aortic aneurysm (Vascular disorders) | 2 | 3
Aortic stenosis (Vascular disorders) | 7 | 1
Aorto-duodenal fistula (Vascular disorders) | 0 | 1
Arterial disorder (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 5 | 5
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Cardiovascular insufficiency (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 14
Diabetic microangiopathy (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 3
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 7
Hypertension (Vascular disorders) | 40 | 48
Hypertensive crisis (Vascular disorders) | 8 | 13
Hypertensive emergency (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 13 | 16
Hypovolaemic shock (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 2
Ischaemia (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Microangiopathy (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 5 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 5
Peripheral ischaemia (Vascular disorders) | 3 | 4
Peripheral vascular disorder (Vascular disorders) | 9 | 13
Phlebitis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 2
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 3
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Varicophlebitis (Vascular disorders) | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 1
Vascular stenosis (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2019) | Darbepoetin Alfa (N=2004)
Anaemia (Blood and lymphatic system disorders) | 102 | 57
Constipation (Gastrointestinal disorders) | 154 | 130
Diarrhoea (Gastrointestinal disorders) | 283 | 279
Nausea (Gastrointestinal disorders) | 227 | 231
Vomiting (Gastrointestinal disorders) | 190 | 200
Asthenia (General disorders) | 166 | 140
Fatigue (General disorders) | 351 | 322
Oedema (General disorders) | 126 | 124
Oedema peripheral (General disorders) | 417 | 414
Bronchitis (Infections and infestations) | 169 | 163
Influenza (Infections and infestations) | 115 | 108
Nasopharyngitis (Infections and infestations) | 179 | 210
Sinusitis (Infections and infestations) | 91 | 112
Upper respiratory tract infection (Infections and infestations) | 182 | 185
Urinary tract infection (Infections and infestations) | 247 | 262
Contusion (Injury, poisoning and procedural complications) | 93 | 111
Fall (Injury, poisoning and procedural complications) | 135 | 165
Blood pressure increased (Investigations) | 102 | 109
Gout (Metabolism and nutrition disorders) | 94 | 106
Hyperglycaemia (Metabolism and nutrition disorders) | 95 | 101
Hyperkalaemia (Metabolism and nutrition disorders) | 106 | 110
Hypoglycaemia (Metabolism and nutrition disorders) | 215 | 225
Arthralgia (Musculoskeletal and connective tissue disorders) | 249 | 257
Back pain (Musculoskeletal and connective tissue disorders) | 266 | 223
Muscle spasms (Musculoskeletal and connective tissue disorders) | 134 | 129
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 117 | 119
Pain in extremity (Musculoskeletal and connective tissue disorders) | 289 | 293
Dizziness (Nervous system disorders) | 206 | 226
Headache (Nervous system disorders) | 161 | 192
Cough (Respiratory, thoracic and mediastinal disorders) | 236 | 214
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 307 | 259
Rash (Skin and subcutaneous tissue disorders) | 80 | 111
Hypertension (Vascular disorders) | 301 | 332
Hypotension (Vascular disorders) | 88 | 110

LIMITATIONS AND CAVEATS:
4047 subjects were enrolled, but before unblinding, all information from 9 subjects was excluded from two sites (3 and 6 subjects, respectively) that did not adhere to Good Clinical Practice guidelines. 4038 subjects were analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.